CLINICAL TRIAL: NCT05583331
Title: Comparison of Two Surgical Sequences "Cataract Surgery Then Vitrectomy" Versus "Vitrectomy Then Cataract Surgery" Under Local-regional Anesthesia. a Pilot, Exploratory, Monocentric, Prospective, Randomized Study
Brief Title: Comparison of Two Surgical Sequences "Cataract Surgery Then Vitrectomy" Versus "Vitrectomy Then Cataract Surgery" Under Local-regional Anesthesia
Acronym: VICAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICAR; 2022-A00886-37 (Other: ANSM)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Cataract; Vitreous Disorder
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Vitrectomy

STUDY DESIGN:
Intervention Model Description: A prospective, randomised, double-arms, parallel, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cataract surgery then Vitrectomy (Active Comparator): Patients will undergo first the cataract surgery then the vitrectomy, as a combined surgery performed on the same day.
  Interventions: Procedure: Cataract surgery; Procedure: Vitrectomy
- Vitrectomy then cataract surgery (Experimental): Patients will undergo first the vitrectomy then the cataract surgery, as a combined surgery performed on the same day.
  Interventions: Procedure: Cataract surgery; Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Cataract surgery — Cataract surgery will be performed as per local practice and standard guidelines.
Procedure: Vitrectomy — Vitrectomy will be performed as per local practice and standard guidelines.

SUMMARY:
Cataracts and vitreo-retinal conditions are frequently associated and can lead to a combined surgery to treat both diseases at the same time. To date, in most cases cataract surgery is usually performed first, then followed by vitrectomy. However, there isn't any standard guidelines indicating what would be the best chronological order, or sequence, when performing those procedures. This randomised, double-arm, open-label study aims at investigating whether the sequence "cataract surgery then vitrectomy" or "vitrectomy then cataract surgery" can have an impact on iris hernia occurence.

DETAILED DESCRIPTION:
Cataracts and vitreo-retinal conditions are frequently associated, such as epimacular membranes, vitreomacular tractions, macular holes, or even macular edema. Cataract is also a frequent complication of posterior vitrectomy. Surgical treatment for pre- or post-vitrectomy cataract is corneal phacoemulsification with intraocular lens implantation.

Many patients undergoing vitrectomy alone consult five to ten years later, without useful vision due to a dense cataract that might be more complicated to treat at a late stage. Indeed, if the phacoemulsification on a previously vitrectomized eye is not an issue in the first years, the intervention can be complicated ten years later, due to nuclear hardness and zonular weakness.

To date, there are no recommendations regarding the surgical sequence for the combination of cataract surgery and vitrectomy. The most-used sequence is to start with cataract surgery and then to perform the vitrectomy most often in 25 gauges (retinal surgery). When we start with cataract surgery under locoregional anesthesia, we often have (in about 15% of cases) iris hernia, which causes intraoperative discomfort (need to put stitches on the cornea), intraoperative miosis, pigments release, which can interfere with visualization during vitrectomy and which require dilating agents use.

The hypothesis of this study is that reversing the order of interventions and starting with vitrectomy could in particular reduce the incidence of intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years old or more
* Patient with macular disease requiring vitrectomy
* Patient with cataract requiring surgery
* Patient suitable for local-regional anesthesia
* Patient suitable for undergoing both surgical procedures consecutively and in any order
* Patient that have given informed consent before performing any study-related procedure
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pseudophakic patients
* Contra-indications to local-regional anesthesia
* Pregnant or breastfeeding patients
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Intraoperative iris hernia occurence | During the combined surgery

SECONDARY OUTCOMES:
Other intraoperative complications occurence | During the combined surgery
Post-operative complications occurence | At 6 months after the combined surgery
Combined surgery duration in minutes | At the end of the combined surgery
Ocular hypertension occurence | At 1 month, 3 months and 6 months after combined surgery
Combined Surgery-related costs assessment | At the time of the combined surgery.
Visual acuity assessment | At 6 months after combined surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Ophtalmique de Somain, Somain, France

IPD SHARING:
Plan to Share IPD: No